CLINICAL TRIAL: NCT03455062
Title: Fertility Study of Women Who Received Organ Transplantation
Acronym: FERTIGREFF
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0092; 2017-A00913-50 (Other: ID-RCB)
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Transplant; Fertility
Keywords: Transplant, fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire about fertility — Recruitment of participants through the list of cardiac, renal, hepatic, pancreatic or pulmonary transplant patients collected from the the Organ Transplant Unit.
  A letter from the the Organ Transplant Unit will initially be sent to patients informing them of the study and if they do not wish to participate they can report their opposition by email.
  A fertility questionnaire will be send and that will have to be returned by the patient in order to be included in the study.
  The questionnaires, anonymous, will be numbered according to their order of return.

SUMMARY:
In terms of immunity, pregnancy can be considered a semi-allogeneic transplant. There are several immunological mechanisms for implantation and maintenance of pregnancy by induction of tolerance without induction of immunosuppression.

This study wants to evaluate the impact of immunodepression on women's fertility by studying the fertility of transplanted cardiac, renal, hepatic and pulmonary women.

DETAILED DESCRIPTION:
A study of HIV-positive immunocompromised patients in medically assisted procreation, published in January 2016, found lower rates of implantation, clinical pregnancy, and newborn babies in these patients compared to HIV-negative patients.

Studying the fertility of transplanted immunocompromised women would provide adequate information on fertility and pregnancy possibilities for these patients, study their fertility on a larger scale and finally better understand the role of immunodepression in fertility.

Pregnancy is considered an allogeneic semi-graft, one can question the fertility of these patients under long-term immunosuppressive treatment. In particular, is there an impact on embryo implantation and on the development of pregnancy? To try to answer this problematic, we propose a retrospective non-interventional study to evaluate the birth rate after spontaneous or induced pregnancy in women who have tried to procreate after transplantation.The data will be collected using questionnaires submitted to the women present in the list of patients transplanted from the Organ Transplant Unit (OTU) of Toulouse University Hospital who have agreed to participate. This will make it possible to retrospectively study fertility data in these patients and to carry out, with the necessary hindsight, statistics on pregnancy rates.

The primary outcome measure: birth rate after spontaneous or induced pregnancy in liver, heart, lung or kidney transplant patients who have attempted to procreate post-transplant is a good primary endpoint because it is a unique clinical criterion. relevant to the purpose of the study, specific and objective.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient who has had a heart, kidney, liver, pancreatic or pulmonary transplant for at least 5 years
* Patients under 40 at the time of transplant
* Patient having given her no opposition to her participation in research

Exclusion Criteria:

* Minor patients
* Patients over 40 at the time of the transplant
* Menopausal patients during organ transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Principal outcome is about the fertility and the pregancy rate
Study Population: Living patients who had a transplant before age 40
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Birth rate | 1 day
  Birth rate after spontaneous or induced pregnancy in women with heart, kidney, liver, pancreatic or pulmonary transplantation

SECONDARY OUTCOMES:
Rates of ectopic pregnancy | 1 day
  Rates of ectopic pregnancy, early or late spontaneous miscarriage, early or late pregnancy, infants born dead, prematurity in women who have tried to procreate post-transplant.
Rates of desire of pregnancy | 1 day
  Rates of desire of pregnancy in these patients and study of the reasons for this lack of desire for pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Jean Parinaud, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No